CLINICAL TRIAL: NCT00040937
Title: A Phase II Trial Of Thalidomide/Dexamethasone Induction Followed By Tandem Melphalan Transplant And Prednisone/Thalidomide Maintenance (A BMT Study)
Brief Title: S0204 Thalidomide, Chemotherapy, and Peripheral Stem Cell Transplant in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0204; S0204 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2002-07-08; First posted 2003-01-27 (Estimated); Results first posted 2013-07-17 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-10

CONDITIONS: Multiple Myeloma
Keywords: stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor; Cyclophosphamide; Dexamethasone; Calcium Dobesilate; Melphalan; Prednisone; Steroids; Thalidomide; Peripheral Blood Stem Cell Transplantation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment arm (Experimental): thalidomide/dexamethasone followed by tandem melphalan peripheral blood stem cell transplantation (with cyclophosphamide and filgrastim or sargramostim support) and prednisone/thalidomide maintenance
  Interventions: Biological: filgrastim; Biological: sargramostim; Drug: cyclophosphamide; Drug: dexamethasone; Drug: melphalan; Drug: prednisone; Drug: thalidomide; Procedure: peripheral blood stem cell transplantation

INTERVENTIONS:
Biological: filgrastim — PBSC collection: 10 mcg/kg SQ days 1-10
  Other Names: G-CSF
Biological: sargramostim — PBSC collection: 500 mcg/m2 SQ day 1 through last apheresis
  1st and 2nd trans: 500 mcg SC or IV days 6-WBC recovery
  Other Names: GM-CSF
Drug: cyclophosphamide — PBSC collection: 1 mg/m2 IV over 45-60 mins day 0
  Other Names: cytoxan
Drug: dexamethasone — 40 mg/d PO days 1-4, 9-12, 17-20
  Other Names: decadron
Drug: melphalan — 1. st trans: 140 mg/m2 IV over 20 mins day -1
  2. nd trans: 200mg/m2 IV over 20 mins day -1
Drug: prednisone — maint: 50 mg/d PO every other day until progression
  Other Names: steroid
Drug: thalidomide — ind: 50 mg increased by 50 mg every week to max 400 mg PO qhs for 35 days maint: 50 mg/d increased by 50 mg every week to 200 mg PO daily until progression
  Other Names: thalomid
Procedure: peripheral blood stem cell transplantation — 2-4 x 10^6/kg IV day 0
  Other Names: stem cell transplant

SUMMARY:
RATIONALE: Thalidomide may stop the growth of cancer cells by stopping blood flow to the cancer. Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell transplant may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells. Giving thalidomide before and after peripheral stem cell transplant may be effective in treating newly diagnosed multiple myeloma.

PURPOSE: This phase II trial is studying how well giving thalidomide with chemotherapy and peripheral stem cell transplant work in treating patients with newly diagnosed multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy and toxicity of thalidomide and dexamethasone as a pre-transplantation induction regimen in patients with multiple myeloma.
* Determine, preliminarily, the safety and efficacy of prednisone and thalidomide maintenance therapy in these patients.
* Correlate chromosome 13 abnormalities with therapeutic response in patients treated with this regimen.
* Correlate specific subsets of chromosome aberrations with event-free and overall survival of patients treated with this regimen.
* Evaluate immune reconstitution and recovery after first and second transplantation in these patients.

OUTLINE: This is a multicenter study.

* Induction chemotherapy: Patients receive oral thalidomide once daily on days 1-35 and oral dexamethasone once daily on days 1-4, 9-12, and 17-20. Treatment repeats every 35 days for 3 courses in the absence of disease progression or unacceptable toxicity.
* Stem cell mobilization and collection: Beginning 5-7 days, but no more than 3 weeks, after completion of induction chemotherapy, patients receive cyclophosphamide IV over 45-60 minutes on day 0, filgrastim (G-CSF) subcutaneously (SC) on days 1-10, and sargramostim (GM-CSF) SC beginning on day 1 and continuing until completion of peripheral blood stem cell (PBSC) collection. Patients begin PBSC collection on day 11 or as soon as blood counts recover.
* First transplantation: Within 3-6 weeks after cyclophosphamide administration, patients receive melphalan IV over 20 minutes on day -1. Patients undergo PBSC infusion on day 0. Patients receive GM-CSF SC or IV beginning on day 6 and continuing until blood counts recover.
* Second transplantation: Between 2-4 months after first transplantation, patients undergo a second tandem melphalan and PBSC transplantation with GM-CSF support as above.
* Maintenance therapy: Beginning 70-90 days post-transplantation, patients receive oral prednisone every other day and oral thalidomide once daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 12 months for 10 years.

PROJECTED ACCRUAL: Approximately 99 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed multiple myeloma requiring treatment

  * Smoldering myeloma with evidence of progressive disease requiring chemotherapy

    * More than 25% increase in M component levels and/or Bence-Jones excretion or symptom development
  * Non-secretory patients with at least 30% bone marrow plasmacytosis
* No IgM peaks unless there is evidence of more than 30% bone marrow plasmacytosis or more than 3 lytic lesions

PATIENT CHARACTERISTICS:

Age

* 18 to 65

Performance status

* Zubrod 0-2 OR
* Zubrod 3-4 based solely on bone pain

Life expectancy

* Not specified

Hematopoietic

* No untreated, unresolved symptomatic hyperviscosity

Hepatic

* Hepatitis B negative

Renal

* Creatinine no greater than 3 mg/dL if in renal failure and on dialysis (after hydration and/or correction of hypercalcemia)

Cardiovascular

* No history of chronic cerebrovascular accident
* No myocardial infarction within the past 6 months
* No unstable angina
* No congestive heart failure that is difficult to control
* No uncontrollable hypertension
* No cardiac arrhythmia that is difficult to control

Pulmonary

* No history of chronic obstructive or chronic restrictive pulmonary disease
* No untreated, unresolved pneumonia
* Pulmonary function tests (PFTs) at least 50% of predicted
* DLCO at least 50% of predicted
* Arterial partial pressure of oxygen greater than 70 if unable to complete PFTs due to bone pain or fracture

Other

* HIV negative
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No untreated, unresolved pathologic fractures
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use at least 2 highly effective methods of contraception for 4 weeks before, during, and for at least 4 weeks after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No more than 8 weeks of prior thalidomide therapy

Chemotherapy

* No prior chemotherapy for this disease

Endocrine therapy

* Prior steroid therapy allowed provided treatment duration was no more than 2 weeks

Radiotherapy

* No prior radiotherapy to more than 50% of the pelvis

Surgery

* Not specified

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2002-06; Primary Completion 2008-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad A. Hussein, MD, Study Chair — The Cleveland Clinic
Locations (141):
- United States (141):
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California Davis Cancer Center, Davis, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Cancer Center, Sacramento, California
  - Piedmont Hospital, Atlanta, Georgia
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Northside Hospital Cancer Center, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - WellStar Cobb Hospital, Austell, Georgia
  - Charles B. Eberhart Cancer Center at DeKalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Kennestone Cancer Center at Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Cancer Research Center of Hawaii, Honolula, Hawaii
  - OnCare Hawaii, Incorporated - Lusitana, Honolulu, Hawaii
  - Queen's Cancer Institute at Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Incorporated, Honolulu, Hawaii
  - OnCare Hawaii, Incorporated - Kuakini, Honolulu, Hawaii
  - St. Francis Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Kapiolani Medical Center at Pali Momi, ‘Aiea, Hawaii
  - St. Luke's Mountain States Tumor Institute - Boise, Boise, Idaho
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - St. Francis Hospital and Health Centers, Beech Grove, Indiana
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Salina Regional Health Center, Salina, Kansas
  - Stormont-Vail Cancer Center, Topeka, Kansas
  - St. Francis Comprehensive Cancer Center, Topeka, Kansas
  - Wesley Medical Center, Wichita, Kansas
  - Louisiana State University Health Sciences Center - Monroe, Monroe, Louisiana
  - Feist-Weiller Cancer Center at Louisiana State University Health Sciences, Shreveport, Louisiana
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Battle Creek Health System Cancer Care Center, Battle Creek, Michigan
  - Bay Regional Medical Center, Bay City, Michigan
  - Mecosta County General Hospital, Big Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - Lacks Cancer Center at Saint Mary's Mercy Medical Center, Grand Rapids, Michigan
  - Spectrum Health Cancer Care - Butterworth Campus, Grand Rapids, Michigan
  - Metropolitan Hospital, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Hackley Hospital, Muskegon, Michigan
  - Northern Michigan Hospital, Petoskey, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Deaconess Billings Clinic - Downtown, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies - Billings, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - St. Vincent Healthcare, Billings, Montana
  - Deaconess Billings Clinic Cancer Center, Billings, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Internal Medicine Associates of Bozeman, Bozeman, Montana
  - St. James Community Hospital, Butte, Montana
  - Big Sky Oncology, Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Sletten Regional Cancer Institute, Great Falls, Montana
  - St. Peter's Hospital, Helena, Montana
  - Glacier Oncology, PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Eastern Montana Cancer Center, Miles City, Montana
  - Community Medical Center, Missoula, Montana
  - Montana Cancer Center at St. Patrick Hospital and Health Sciences Center, Missoula, Montana
  - Montana Cancer Specialists at Montana Cancer Center, Missoula, Montana
  - Judy L. Schmidt, MD, FACP, P. C., Missoula, Montana
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina
  - McDowell Cancer Center at Akron General Medical Center, Akron, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Riverside Methodist Hospital Cancer Care, Columbus, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Grant Riverside Cancer Services, Columbus, Ohio
  - Mount Carmel West Hospital, Columbus, Ohio
  - Doctors Hospital at Ohio Health, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital, Dayton, Ohio
  - David L. Rike Cancer Center at Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Cancer Care Center, Dayton, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Charles F. Kettering Memorial Hospital, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - MedCentral - Mansfield Hospital, Mansfield, Ohio
  - Strecker Cancer Center at Marietta Memorial Hospital, Marietta, Ohio
  - Middletown Regional Hospital, Middletown, Ohio
  - Licking Memorial Cancer Care Program at Licking Memorial Hospital, Newark, Ohio
  - Mercy Medical Center Oncology Unit, Springfield, Ohio
  - Community Hospital of Springfield and Clark County, Springfield, Ohio
  - UVMC Cancer Care Center at Upper Valley Medical Center, Troy, Ohio
  - Mount Carmel Cancer Services at Mount Carmel St. Ann's Hospital, Westerville, Ohio
  - United States Air Force Medical Center Wright-Patterson, Wright-Patterson AFB, Ohio
  - Ruth G. McMillan Cancer Center at Greene Memorial Hospital, Xenia, Ohio
  - Genesis - Good Samaritan Hospital, Zanesville, Ohio
  - Legacy Mount Hood Medical Center, Glesham, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Comprehensive Cancer Center at Legacy Good Samaritan Hospital & Medical Center, Portland, Oregon
  - Providence Cancer Center at Providence Portland Medical Center, Portland, Oregon
  - CCOP - Columbia River Oncology Program, Portland, Oregon
  - Providence St. Vincent Medical Center, Portland, Oregon
  - Institute of Oncology at Vilnius University, Portland, Oregon
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Rose Ramer Cancer Clinic at Anderson Area Medical Center, Anderson, South Carolina
  - Bon Secours St. Francis Health System, Greenville, South Carolina
  - Greenville Hospital System Cancer Center, Greenville, South Carolina
  - CCOP - Greenville, Greenville, South Carolina
  - Gibbs Regional Cancer Center at Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Wilford Hall Medical Center, Lackland Air Force Base, Texas
  - UMC Southwest Cancer and Research Center, Lubbock, Texas
  - Auburn Regional Center for Cancer Care, Auburn, Washington
  - St. Joseph Hospital Community Cancer Center, Bellingham, Washington
  - Olympic Hematology and Oncology, Bremerton, Washington
  - Regional Cancer Center at Providence Hospital, Centralia, Washington
  - St. Francis Hospital, Federal Way, Washington
  - Skagit Valley Hospital Cancer Care Center, Mount Vernon, Washington
  - Providence St. Peter Hospital Regional Cancer Center, Olympia, Washington
  - Capital Medical Center, Olympia, Washington
  - Good Samaritan Cancer Center, Puyallup, Washington
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Group Health Central Hospital, Seattle, Washington
  - Harborview Medical Center, Seattle, Washington
  - Swedish Cancer Institute at Swedish Medical Center - First Hill Campus, Seattle, Washington
  - University Cancer Center at University of Washington Medical Center, Seattle, Washington
  - North Puget Oncology at United General Hospital, Sedro-Woolley, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Allenmore Hospital, Tacoma, Washington
  - CCOP - Northwest, Tacoma, Washington
  - St. Joseph Medical Center at Franciscan Health System, Tacoma, Washington
  - St. Clare Hospital, Tacoma, Washington
  - Southwest Washington Medical Center Cancer Center, Vancouver, Washington
  - Central Washington Hospital, Wenatchee, Washington
  - Wenatchee Valley Clinic, Wenatchee, Washington
  - Community Comprehensive Cancer Center at Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Welch Cancer Center, Sheridan, Wyoming

REFERENCES:
- [Result] Hussein MA, Bolejack V, Zonder JA, Durie BG, Jakubowiak AJ, Crowley JJ, Barlogie B. Phase II study of thalidomide plus dexamethasone induction followed by tandem melphalan-based autotransplantation and thalidomide-plus-prednisone maintenance for untreated multiple myeloma: a southwest oncology group trial (S0204). J Clin Oncol. 2009 Jul 20;27(21):3510-7. doi: 10.1200/JCO.2008.19.9240. Epub 2009 Jun 22. PMID 19546405
- [Result] Hussein MA, Jakubowiak AJ, Bolejack V, et al.: S0204: melphalan (MEL)-based tandem autotransplants (TAT) for multiple myeloma (MM) with thalidomide/dexamethasone (TD) induction and thalidomide/prednisone (TP) maintenance: a phase II trial of the Southwest Oncology Group. [Abstract] Blood 108 (11): A-3088, 2006.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at participating cooperative group institutions.
Period: Induction/PBSC Mobilization
Arm/Group | Treatment Arm
Started | 147 (147 registered to this period; 142 were eligible and analyzable; 140 were assessable for toxicity.)
Completed | 110
Not Completed | 37
Period: Autologous PBSCT
Arm/Group | Treatment Arm
Started | 108 (108 registered to this period; 105 were eligible and analyzable; 105 were assessable for toxicity.)
Completed | 77
Not Completed | 31
Period: Maintenance
Arm/Group | Treatment Arm
Started | 76
Completed | 76 (Patients remained on protocol therapy until progression.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Arm
Number analyzed (Participants) | 142
Age, Continuous [Median (Full Range); unit: years] | 57 (23-66) [23 to 66]
Gender [Count of Participants; unit: Participants]
  Female | 56
  Male | 86
Region of Enrollment [Number; unit: participants]
  United States | 142

OUTCOME MEASURES:

1. Secondary Outcome: Assess Toxicity of Thalidomide/Dexamethasone as a Pre-transplant Induction Regimen.
Description: To assess Grade 3-5 AE related to thalidomide/dexamethasone when administered as a pre-transplant induction regimen.
Time Frame: Induction
Population: All participants receiving at least one dose of induction therapy
Measure: Number; unit: Participants
Arm/Group | Induction/PBSC Mobilization
Number analyzed (Participants) | 140
Participants | 2

2. Primary Outcome: Overall Survival
Time Frame: 4-7 years
Measure: Number (95% Confidence Interval); unit: proportion surviving at 4 years
Arm/Group | Treatment Arm
Number analyzed (Participants) | 142
proportion surviving at 4 years | .64 [.55 to .74]
Statistical Analysis 1: Comparison: Treatment Arm; The study was designed to have 82% power for detecting a 50% improvement in survival from a median of 4 years, as observed in SWOG S9321; Test type: Superiority or Other; Kaplan and Meier; 4-yr survival (%) = 64, 95% CI 2-sided [55 to 74]

ADVERSE EVENTS:
Time Frame: Report through 4/10/2007 to match data reported in MS.
Arm/Group | Induction/PBSC Mobilization | Autologous PBSCT | Prednisone + Thalidomide
Serious Adverse Events (participants affected / at risk) | 7/140 | 0/105 | 1/76
Other Adverse Events (participants affected / at risk) | 140/140 | 105/105 | 74/76
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction/PBSC Mobilization (N=140) | Autologous PBSCT (N=105) | Prednisone + Thalidomide (N=76)
Supraventricular arrhythmia (Cardiac disorders) | 2 | 0 | 0
GI-other (Gastrointestinal disorders) | 1 | 0 | 0
Respiratory infect w/ neutrop (Infections and infestations) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Apnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Thrombosis/embolism (Vascular disorders) | 2 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction/PBSC Mobilization (N=140) | Autologous PBSCT (N=105) | Prednisone + Thalidomide (N=76)
Anemia (Blood and lymphatic system disorders) | 73 | 94 | 23
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 64 | 0
Transplant-pRBC transfusion (Blood and lymphatic system disorders) | 0 | 7 | 0
Transplant-plt transfusion (Blood and lymphatic system disorders) | 0 | 6 | 0
Arrhythmia, NOS (Cardiac disorders) | 0 | 7 | 0
Palpitations (Cardiac disorders) | 7 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 5
Sinus tachycardia (Cardiac disorders) | 0 | 6 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 5
Cushingoid appearance (Endocrine disorders) | 12 | 0 | 5
Blurred vision (Eye disorders) | 14 | 0 | 5
Cataract (Eye disorders) | 0 | 0 | 4
Dry eye (Eye disorders) | 0 | 0 | 5
Abdominal pain/cramping (Gastrointestinal disorders) | 7 | 15 | 4
Constipation/bowel obstruction (Gastrointestinal disorders) | 85 | 17 | 35
Diarrhea without colostomy (Gastrointestinal disorders) | 21 | 84 | 12
Dyspepsia/heartburn (Gastrointestinal disorders) | 19 | 28 | 13
Esophagitis/dysphagia (Gastrointestinal disorders) | 0 | 40 | 0
GI Mucositis, NOS (Gastrointestinal disorders) | 0 | 7 | 0
GI-other (Gastrointestinal disorders) | 0 | 6 | 4
Mouth dryness (Gastrointestinal disorders) | 8 | 9 | 8
Nausea (Gastrointestinal disorders) | 54 | 96 | 9
Stomatitis/pharyngitis (Gastrointestinal disorders) | 9 | 76 | 0
Vomiting (Gastrointestinal disorders) | 24 | 68 | 7
Edema (General disorders) | 61 | 50 | 24
Fatigue/malaise/lethargy (General disorders) | 114 | 92 | 52
Fever without neutropenia (General disorders) | 38 | 56 | 12
Pain-other (General disorders) | 22 | 17 | 22
Rigors/chills (General disorders) | 18 | 36 | 0
Sweating (General disorders) | 16 | 0 | 0
Allergic reaction (Immune system disorders) | 0 | 6 | 0
Infection w/o 3-4 neutropenia (Infections and infestations) | 38 | 14 | 36
Infection with 3-4 neutropenia (Infections and infestations) | 0 | 19 | 0
Respiratory infection, unk ANC (Infections and infestations) | 0 | 0 | 4
Local injection site reaction (Injury, poisoning and procedural complications) | 7 | 0 | 0
Alkaline phosphatase increase (Investigations) | 19 | 13 | 4
Bilirubin increase (Investigations) | 7 | 13 | 0
Creatinine increase (Investigations) | 16 | 19 | 12
Hypercholesterolemia (Investigations) | 0 | 0 | 5
Leukopenia (Investigations) | 36 | 90 | 26
Lymphopenia (Investigations) | 0 | 14 | 10
Neutropenia/granulocytopenia (Investigations) | 25 | 97 | 14
SGOT (AST) increase (Investigations) | 16 | 15 | 16
SGPT (ALT) increase (Investigations) | 25 | 16 | 18
Thrombocytopenia (Investigations) | 52 | 91 | 9
Transplant-thrombocytopenia (Investigations) | 0 | 6 | 0
Weight gain (Investigations) | 21 | 0 | 24
Weight loss (Investigations) | 9 | 12 | 4
Anorexia (Metabolism and nutrition disorders) | 26 | 50 | 4
Dehydration (Metabolism and nutrition disorders) | 7 | 7 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 7 | 0 | 6
Hyperglycemia (Metabolism and nutrition disorders) | 69 | 34 | 39
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 9 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 4
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 7 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 25 | 35 | 5
Hypocalcemia (Metabolism and nutrition disorders) | 45 | 42 | 15
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 7 | 6
Hypokalemia (Metabolism and nutrition disorders) | 30 | 34 | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 14 | 21 | 0
Hyponatremia (Metabolism and nutrition disorders) | 14 | 23 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 17 | 4
Metabolic-other (Metabolism and nutrition disorders) | 0 | 0 | 9
Arthralgia (Musculoskeletal and connective tissue disorders) | 16 | 6 | 13
Bone pain (Musculoskeletal and connective tissue disorders) | 73 | 41 | 29
Chest pain,not cardio or pleur (Musculoskeletal and connective tissue disorders) | 9 | 6 | 4
Joint,muscle,bone-other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 9
Muscle weakness (not neuro) (Musculoskeletal and connective tissue disorders) | 10 | 0 | 8
Myalgia (Musculoskeletal and connective tissue disorders) | 29 | 16 | 10
Myalgia/arthralgia, NOS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4
Ataxia (incoordination) (Nervous system disorders) | 0 | 0 | 4
Dizziness/light headedness (Nervous system disorders) | 39 | 23 | 19
Headache (Nervous system disorders) | 20 | 35 | 10
Memory loss (Nervous system disorders) | 0 | 0 | 5
Neuro-other (Nervous system disorders) | 8 | 0 | 6
Neuropathic pain (Nervous system disorders) | 0 | 0 | 5
Sensory neuropathy (Nervous system disorders) | 83 | 16 | 60
Somnolence/consciousness loss (Nervous system disorders) | 15 | 0 | 9
Taste disturbance (Nervous system disorders) | 14 | 8 | 0
Tremor (Nervous system disorders) | 20 | 0 | 9
Weakness (motor neuropathy) (Nervous system disorders) | 17 | 0 | 16
Anxiety/agitation (Psychiatric disorders) | 21 | 22 | 13
Confusion (Psychiatric disorders) | 0 | 0 | 5
Depression (Psychiatric disorders) | 19 | 10 | 18
Insomnia (Psychiatric disorders) | 28 | 20 | 15
Personality/behavioral change (Psychiatric disorders) | 12 | 0 | 4
Sexual/reproductive-other (Reproductive system and breast disorders) | 0 | 0 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 27 | 18
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 39 | 25 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 0
Hiccoughs (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 8 | 0 | 0
Lung-other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4
Pleural effusions (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 0
Pneumonitis/infiltrates (Respiratory, thoracic and mediastinal disorders) | 7 | 0 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 9 | 35 | 0
Eryth/rash/eruption/desq, NOS (Skin and subcutaneous tissue disorders) | 0 | 0 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 9 | 16 | 6
Rash/desquamation (Skin and subcutaneous tissue disorders) | 42 | 35 | 10
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 0 | 6
Hot flashes (Vascular disorders) | 0 | 0 | 5
Hypertension (Vascular disorders) | 0 | 9 | 9
Hypotension (Vascular disorders) | 21 | 27 | 4
Thrombosis/embolism (Vascular disorders) | 17 | 7 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No